CLINICAL TRIAL: NCT00449943
Title: Comparison of Cardiac Computed Tomographic Angiography (CTA) to Tc-99m Single Photon Emission Computed Tomography (SPECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Benjamin Chow, MD, Ottawa Heart Institute Research Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2006360-01H
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac Invasive Catheterization Angiography; Single Photon Emission Computed Tomography; Computed Tomography Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: Computed Tomographic Angiography — CT scan
Procedure: Myocardial Perfusion Imaging Scan — SPECT

SUMMARY:
Cardiovascular disease and ischemic heart disease is the #1 killer in Canada. Currently, Cardiac invasive catheterization angiography (CICA) is the gold standard for the assessment of the arteries in the heart. However, cardiac catheterization has risks which prohibit its use in all patients. These risks include: death, heart attack, stroke and bleeding. Cardiac computed tomography angiography (CTA) is a new non-invasive technology which may enable the evaluation of patients' coronary anatomy without exposing patients to the risks of invasive cardiac catheterization.

The purpose of this project is to compare CT angiography (CTA) to Tc-99m single photon emission computed tomography (Tc-99m SPECT)

We will enroll patients who are waiting for a CICA or who have been referred for a TC-99m SPECT or CTA scans at the University of Ottawa Heart Institute. Consenting patients who are waiting for a CICA will have both a CTA and a Tc-99m SPECT scan. Consenting patients referred for a CTA or Tc-99m SPECT will have both the CTA and Tc-99m SPECT in a random order but not CICA (unless ordered by your physician).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for Tc-99m SPECT or CTA; or
* Patients referred for CICA without preceding (< 12 months) MPI or CTA

Exclusion Criteria:

* Previous revascularization (PCI or CABG)
* Age < 18 years or lack of consent
* Renal Insufficiency (GFR < 60 ml/min)
* Allergy or contraindication to contrast agent or dipyridamole
* Refractory angina requiring urgent/emergent coronary angiography
* Contraindication to radiation exposure (e.g. pregnancy)
* Uncontrolled HR
* Atrial fibrillation, frequent atrial or ventricular ectopy (> 1/minute)
* Unable to perform 10 second breath-hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To measure the accuracy of CTA to SPECT for the diagnosis of CAD | 1 year

SECONDARY OUTCOMES:
To examine the accuracy of CTA predicting the mode of treatment: Medical therapy or revascularization (PCI versus CABG) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin JW Chow, MD, FRCPC, Principal Investigator — Ottawa Heart Institute Research Corporation; Robert Beanlands, MD, Study Chair — Ottawa Heart Institute Research Corporation; Terrence Ruddy, MD, Study Chair — Univeristy of Ottawa Heart Institute; Carole Dennie, MD, Study Chair — The Ottawa Hospital
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- See also: University of Ottawa Heart Institute — http://www.ottawaheart.ca